CLINICAL TRIAL: NCT01018498
Title: Pilot Study Using a Dietary Intervention for Children With Irritable Bowel Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: American College of Gastroenterology (Other); Texas Medical Center Digestive Disease Center (Unknown); NASPGHAN Foundation (Other Government)
Responsible Party: Principal Investigator, Bruno Chumpitazi, Assistant Professor, Baylor College of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-25005
Record Dates: First submitted 2009-10-28; First posted 2009-11-23 (Estimated); Last update posted 2018-01-18 (Actual); Status verified 2018-01

CONDITIONS: Irritable Bowel Syndrome
Keywords: Irritable Bowel Syndrome; Children
MeSH Terms: conditions — Irritable Bowel Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Restricted FODMAPs diet (Experimental): Restricted fermentable substrate diet for 1 week
  Interventions: Behavioral: Restricted FODMAPs diet

INTERVENTIONS:
Behavioral: Restricted FODMAPs diet — Restricted fermentable substrate diet

SUMMARY:
Malabsorption of certain foods (e.g. lactose) has been proposed as a cause of irritable bowel syndrome in adults and children. Recently, a diet that lowers intake of a combination of foods has been found to be effective in adults with IBS identified with fructose malabsorption.

The purpose of this study is to determine whether a restricted fermentable substrate diet is effective in the treatment of irritable bowel syndrome in children.

DETAILED DESCRIPTION:
Up to 19% of school-aged children have recurrent abdominal pain (RAP), accounting for 5% of all pediatric office visits and increased morbidity. The majority of children with RAP have irritable bowel syndrome (IBS) with up to 60% these children going on to develop IBS as adults. IBS accounts for up to 8 billion dollars a year of healthcare costs in adults within the United States. Successful interventions that ameliorate symptoms in childhood IBS may have an impact into adulthood, however current clinical interventions are often ineffective.

As in adults, the etiology of childhood IBS is multi-factorial, with food intolerance and increased gastrointestinal inflammation being potential factors. Another factor, that of malabsorption of fermentable substrates (e.g., fructose), has frequently been postulated as a form of food intolerance that exacerbates IBS symptoms in adults and children. Studies suggest up to 61% of children with RAP have fructose malabsorption. The interactions between factors such as increased gastrointestinal inflammation and malabsorption of fermentable substrates and they relate to an individual patient is currently unknown.

Recently, a diet that lowers intake of a combination of foods has been found to be effective in adults with IBS identified with fructose malabsorption. This diet has not been used in children with IBS nor has its mechanism(s) of efficacy been explored. This pilot project focuses on using a restricted fermentable substrate diet as a treatment in children with IBS, while evaluating decreased bacterial fermentation gas production and decreased gastrointestinal inflammation as mechanisms of its effect.

Using a prospective, open label design in children meeting Rome III childhood IBS criteria, our Specific Aims are to: 1) Characterize the effectiveness of a restricted FODMAPs diet in improving symptoms (number of abdominal pain episodes; primary endpoint); 2) To determine the mechanisms by which a restricted FODMAPs diet may work. We Hypothesize that: 1) A restricted FODMAPs diet will improve abdominal pain symptoms associated with childhood IBS and identified fructose malabsorption; 2) A restricted FODMAPs diet will improve symptoms in part by decreasing bacterial fermentation gas production amongst other potential mechanisms.

The results of this proposal may, if applied on a larger scale, aid a large number of children with IBS and potentially provide insight into the mechanism(s) behind successful dietary interventions for childhood IBS.

ELIGIBILITY:
Inclusion Criteria:

* Ages 7-17 years
* Meet criteria for Rome III irritable bowel syndrome
* Negative physician evaluation within past year for abdominal pain

Exclusion Criteria:

* Diabetes or other problem requiring specialized diet
* Red dye allergy
* Unable to eat by mouth
* Malnutrition or recent rapid weight loss
* Psychotherapy for abdominal pain
* Significant cognitive impairment or psychiatric co-morbidity
* Frequent vomiting
* History of suicide attempt
* Non-English speaking parent or child
* Chronic medical condition (excluding asthma)
* Antibiotic usage, medicinal probiotic usage, or neuromodulator (e.g. amitriptyline) usage within the past 3 months
* Start of or change in gastrointestinal medication (e.g. laxative) that may cause or ameliorate symptoms within the past month

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 12 (Actual)
Dates: Start 2009-10; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Improvement in pain frequency | Prior to and after 1 week of treatment

SECONDARY OUTCOMES:
Changes in GI Transit Time | Prior to and after 1 week of treatment
Changes in Breath Hydrogen and Methane production | Prior to and after 1 week of treatment
Changes in GI Permeability | Prior to and after 1 week of treatment
Changes in fecal microbiome | Prior to and after 1 week of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Bruno P Chumpitazi, M.D., M.P.H., Principal Investigator — Baylor College of Medicine
Locations (2):
- United States (2):
  - Children's Nutrition Research Center, Houston, Texas
  - Texas Children's Hospital, Houston, Texas

REFERENCES:
- [Result] Chumpitazi BP, Hollister EB, Oezguen N, Tsai CM, McMeans AR, Luna RA, Savidge TC, Versalovic J, Shulman RJ. Gut microbiota influences low fermentable substrate diet efficacy in children with irritable bowel syndrome. Gut Microbes. 2014 Mar-Apr;5(2):165-75. doi: 10.4161/gmic.27923. Epub 2014 Jan 27. PMID 24637601